CLINICAL TRIAL: NCT04647617
Title: Effects of 12- Weeks of Quantitative Weight-bearing Progressive Resistance Exercise Training on Glycemia Control and Improving Muscle Strength With Type 2 Diabetes Combine Pre-sarcopenia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu- Hsuan Chien (Other)
Responsible Party: Sponsor-Investigator, Yu- Hsuan Chien, Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202001276B0
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Twelve Week Quantitative Weight Bearing of Resistance Training Effect on Glycemic Control and Muscle Strength
Keywords: Resistance training；Muscle strength；Glycemic control

STUDY DESIGN:
Intervention Model Description: Forty adult diagnosis with T2DM with pre-sarcopenia patient randomly assigned to experimental group and control group. Experimental group wearing 0.5 kg quantitative sandbag 12~15 Repetitions/set X 5 set X 3day.control group keep normal lives
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quantitative Weight-bearing (Experimental): Experimental wearing 0.5 kg quantitative sandbag 12~15 Repetitions/set X 5 set X 3day. Weight adjustment: After the first month of intervention, if the experimental can perform for more than 20 repetitions/set , we will asked to increase the weight of the sandbag to 1 kg until the end of the experiment
  Interventions: Behavioral: Quantitative weight -bearing and report exercise sign data every weekly
- Control group (Placebo Comparator): They are keep their normal live style
  Interventions: Behavioral: Quantitative weight -bearing and report exercise sign data every weekly

INTERVENTIONS:
Behavioral: Quantitative weight -bearing and report exercise sign data every weekly — keep their normal live style
  Other Names: Self-manage

SUMMARY:
According to the International Diabetes Federation (IDF) in 2017 investigator found that the incidence of type 2 diabetes is currently 425 million people aged 20 to 79 in the world, and this data will increase o 629 million at 2045, The etiology of more than 90% is related to aging, it has become a serious challenge to public health.

Sarcopenia is a newly noticed severe syndrome characterized by reduced walking speed, decreased grip strength, and decreased muscle mass. Patients with type 2 diabetes are at risk of sarcopenia and are those with normal blood sugar. One of the main ways to improve the face of sarcopenia is to exercise intensity. By carrying out a gradual training plan instead of using different weights, it will lead to muscle hypertrophy and increase in muscle strength to achieve muscle gain. In view of the fact that the commercially available sandbags are cheap and easy to obtain, the weight is fixed, and the use variability is high, it is expected to introduce quantitative weight-bearing progressive exercises in type 2 diabetes and have symptoms of muscle loss to improve muscle mass, and to control blood sugar. The quality of life can have better benefits.

DETAILED DESCRIPTION:
Purpose:This study aim is effectiveness of 12 weeks quantitative weight-bearing progressive exercise training in patients with type 2 diabetes mellitus(T2DM) with pre-sarcopenia promotion muscle strength and blood sugar control.

Hypothesis:After 12 weeks of quantitative sandbag training , the experimental group can have a significant increase in the muscle mass of the upper and lower limbs、grip strength、5-time chair stand test、Lipid profile、glycemic control(HbA1c) and quality of life.

Methods:This study will be a randomized controlled trial. Forty adult diagnosis with T2DM with pre-sarcopenia patient randomly assigned to experimental group and control group. Experimental group wearing 0.5 kg quantitative sandbag 12~15 Repetitions/set X 5 set X 3day. Weight adjustment: After the first month of intervention, if the experimental can perform for more than 20 repetitions/set , we will asked to increase the weight of the sandbag to 1 kg until the end of the experiment Conditions:The effectiveness of 12 weeks quantitative weight-bearing can improvement of Glycemic control and limb muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 ~80 years
* T2DM
* Physician and check Calf circumference (M: <34 cm, F: <33 cm)、handgrip strength (M: <28 kg, F: <18 kg)

Exclusion Criteria:

* Inability to perform any self -activity
* DM with lower limb neuropathy, r
* DM with Retinopathy
* Stroke
* Foot opening wound
* Past history even doing limb resistance training;
* Easy fall down high risk patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c level | up to 12 week of invention
  follow blood glucose control
muscle strength | up to 12 weeks of intervention
  follow hand grip male.If the hand grip show weakness it mean the worse of muscle strength
muscle mass | up to 12 weeks of invention
  Use BIA(Bioelectrical impedance analysis)follow muscle mass,
5-time chair stand test | up to 12 weeks of invention
  follow low limb muscle strength .The higher number of seconds, it mean the worse the lower limb ability

SECONDARY OUTCOMES:
WHOQOL-BREF World Health Organization Quality of Life Taiwan version | up to 12 week of invention
  follow T2DM with pre-sarcopenia quality of life. The Questionnaire include four domain: psychological domain, social domain, environment domain and Taiwan local domain.This questionnaire scale higher is more better
  follow T2DM with pre-sarcopenia

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jen Tsai, Study Director — Kaohsiung Chang Gung Medication Hosipital
Locations (1):
- Yu-Hsuan Chien, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage, and then share with other researchers after publication